CLINICAL TRIAL: NCT00142272
Title: Randomised, Open, Parallel Group Clinical Trial to Compare the Efficacy and Safety of a Single Dose of Ciprofloxacin Oral Suspension 20 mg/kg With a 3-day Course of Erythromycin Oral Suspension Administered in a Dose of 12.5 mg/kg Every 6 Hours (12 Doses) in the Treatment of Children,With Clinically Severe Cholera Due to V. Cholerae O1 or O139.
Brief Title: Single Dose Ciprofloxacin in the Treatment of Childhood Cholera:Randomized Controlled Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Bayer (Industry); NEMC (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000-032_
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2005-09

CONDITIONS: Cholera
Keywords: Ciprofloxacin; children; V.cholerae O1 and O139; drug resistance; Bangladesh
MeSH Terms: conditions — Cholera | interventions — Ciprofloxacin

INTERVENTIONS:
Drug: Ciprofloxacin

SUMMARY:
The study will be conducted to compare the efficacy and safety of a single dose of ciprofloxacin oral suspension 20 mg/kg with a 3-day course of erythromycin oral suspension administered in a dose of 12.5 mg/kg every 6 hours (12 doses) in the treatment of children, aged 2-15 years with clinically severe cholera due to V. cholerae O1 or O139.

We hypothesize that single dose ciprofloxacin would result in similar outcome in the clinicalcurewith that of erythromycin given in multiple doses.

DETAILED DESCRIPTION:
Eligible patients will be admitted to the Clinical Study Ward of the Dhaka and Matlab Hospitals of ICDDR,B. Upon admission, their weight (dehydrated weight) and vital signs will be recorded, and a thorough physical examination, including assessment of dehydration (following WHO guidelines), will be made. Patients will then be rehydrated using intravenous Dhaka Solution (133, 13, 98 and 48 mmol/l of sodium, potassium, chloride and bicarbonate, respectively) over 3-4 hours. Thereafter, they will be observed over a 4-hour Observation Period when their hydration will be maintained using the rice-based oral rehydration solution (ORS) (containing 3.5, 2.5, 1.5 and 50 gram/l of sodium chloride, sodium bicarbonate, potassium chloride and rice powder). Dhaka Solution, as used for initial rehydration, will be used for patients whose hydration cannot be maintained by rice-based ORS.Patients who have a stool output of 20 ml/kg or more during the Observation Period, and who have V. cholerae demonstrated in dark-field microscopic examination of their freshly passed stool sample, will be enrolled upon obtaining written informed consent of their parents or guardians. If possible, assent must be obtained from the child. Patients will then be randomly assigned to receive one of the two treatment regimens. Children will be hospitalised for 5 days, from the initiation of study drug or until resolution of their diarrhoea, whichever will be longer, and they will be asked to return for a follow-up evaluation 10 to 14 days after study entry. Patients are to return for a further follow-up visit at 4 to 6 weeks (Day 28 to Day 42).Patients who develop joint changes during therapy, or during the follow-up period, must be followed up. Any new objective finding noted on clinical joint or gait assessment will be thoroughly evaluated by the investigator. This evaluation may include diagnostic procedures, such as MRI and/or joint fluid assessments, as appropriate. Patients with joint changes during therapy, or during the follow-up period, should be followed up until:a) The adverse event has been resolved orb) Until further change in the patient's condition is unlikely and a final causality assessment has been made. This may be shorter or longer than 3 months from the time of discharge.Medical history will be obtained and a thorough physical examination will be performed daily. Vital signs and intake/output records will be maintained as from the initiation of rehydration.Patients will be closely monitored through bacteriological and laboratory assessments. Blood, urine and stool specimens will be taken at various time points. Stool culture for enteric pathogens will be done before initiation of the study drug, on study Day 3 and at follow-up visits. Rectal swab culture for V. cholerae will be done on each day of the study during the hospitalisation period, and at follow-up (10 to 14 days and 4 to 6 weeks). Complete blood count, serum electrolytes and creatinine, total bilirubin, SGPT and alkaline phosphatase will be determined before initiation of study drug and on study Day 5. (If the baseline creatinine is > 200 mcmol/L, creatinine will also be determined 24 hours post-administration of first dose of study medication, and any patient with a creatinine > than 200 mcmol/L will be considered as suffering from renal failure and will be withdrawn from the trial.) If possible, urinalysis will be done before initiation of drug therapy and on Day 5 of the study. Serum concentration of ciprofloxacin will be determined on the first day of the study at various time intervals after the first dose of the study drug.

ELIGIBILITY:
Inclusion Criteria:

Age: 2-15 years. Gender: male. Duration of illness: <24 hours. Written informed consent for participation in the study from either of the parents, or guardian, and oral assent from children aged ³ 8 years.

Severe dehydration according to World Health Organisation (WHO) guidelines. Positive stool dark field microscopic examination for V. cholerae.

Exclusion Criteria:

History of receiving any antimicrobial agent (including study drugs) effective in the treatment of V. cholerae within 72 hours of screening.

Concomitant infection(s) requiring antimicrobial therapy. A concomitant illness that may interfere with the evaluation of outcome or safety of the study drugs.

Patients with known chronic renal insufficiency. [As all cholera patients with moderate to severe dehydration have pre-renal insufficiency on admission, and as it is not possible to detect whether a patient has renal failure until the patient has been hydrated for at least 24 hours, serum creatinine will be checked 24 hours post-administration of first dose of study medication, on Day 5, and at any time as clinically indicated. (If the baseline creatinine is > 200 mcmol/L, any patient with creatinine > than 200 mcmol/L 24 hours post-administration, will be considered as suffering from renal failure and will be withdrawn from the trial.) Patients with known cardiac or hepatic impairment, i.e. SGOT/SGPT or bilirubin > 3 times the upper limit of normal, and patients with a history of central nervous system (CNS) disorders (known risk of experiencing seizures, a history of convulsive disorders or head injury trauma, currently on anti-seizure medication or within two months post-stroke).

Patients previously enrolled in the study. Patients participating in any clinical study within one month prior to study entry.

Patients' known to have AIDS. Patients treated with quinolones in the 14 days prior to the study. Patients known to have underlying rheumatological disease, joint problems, etc. Patients with a known hypersensitivity to any of the study drug regimens or related compounds (including fluoroquinolones and macrolides).

Female patients who are lactating, or are sexually active and using unreliable contraception.

Patients having a known underlying rheumatological disease, joint problems secondary to trauma or pre-existing conditions known to be associated with arthropathy.

Patients with conditions precluding the performance of a reliable series of musculoskeletal examinations are to be excluded from trial participation.

Ages: 2 Years to 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180
Dates: Start 2001-05; Study Completion 2002-07

PRIMARY OUTCOMES:
Rates of clinical success

SECONDARY OUTCOMES:
Rates of bacteriologic success at test of cure visit.
Duration of diarrhoea.
Rates of clinical relapse.
Rates of bacteriologic relapse.
Duration of faecal excretion of V. cholerae O1 or V. cholerae O139.
Measurements of six-hourly volume of watery stool will be done for the period in which patients are hospitalised.
Proportion of patients requiring unscheduled intravenous fluids.
Frequency of vomiting and its volume.
Frequency of stool per day.
Frequency of vomit per day.
Safety.
PK-assessment of serum and stool.

CONTACTS AND LOCATIONS:
Overall Officials: Debasish Saha, MBBS,MS, Study Director — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

REFERENCES:
- [Derived] Saha D, Khan WA, Karim MM, Chowdhury HR, Salam MA, Bennish ML. Single-dose ciprofloxacin versus 12-dose erythromycin for childhood cholera: a randomised controlled trial. Lancet. 2005 Sep 24-30;366(9491):1085-93. doi: 10.1016/S0140-6736(05)67290-X. PMID 16182896